CLINICAL TRIAL: NCT03487796
Title: MySTYLE: Online Family-based HIV Prevention for Non-heterosexual Black Adolescent Males in the South
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Larry K. Brown, Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH113384 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-04-04 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Hiv; Adolescent Behavior; Family Relations; Sexual Orientation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Adolescent Behavior; Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MySTYLE (Experimental): MySTYLE is online, brief and encourages parent-adolescent communication about sex and HIV prevention. Participants (non-heterosexual Black adolescent males and parents/caregivers) will receive two texts per week (for eight weeks) with links to intervention content that includes video, games and graphics to improve knowledge, motivation and skills for HIV prevention. Topics include assertive communication, sexual safety, goal setting, and resilience.
  Interventions: Behavioral: MySTYLE
- Waitlist Control (Other): Participants randomized to the waitlist control will be eligible to receive the eight-week MySTYLE intervention after the completion of the 4-month follow-up assessment. During their first four months of participation, waitlist control participants will not receive any intervention materials.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: MySTYLE — Youth and parents will receive two secure texts or emails to their cell phone or preferred device weekly (for eight weeks). Each text/email will contain a link to new media content designed to (1) improve sexual health knowledge surrounding HIV/AIDs and sexually transmitted infections, (2) increase acceptance of young Black men of all backgrounds (sexual, economic, and family), and (3) improve parent and adolescent relationships and communication.
  Arms: MySTYLE
Other: Waitlist Control — Youth and parents will not receive intervention materials for the first four months of participation. At the completion of the 4-month follow-up assessment, youth and parents will be eligible to receive two secure texts or emails to their cell phone or preferred device weekly (for eight weeks). Each text/email will contain a link to new media content designed to (1) improve sexual health knowledge surrounding HIV/AIDs and sexually transmitted infections, (2) increase acceptance of young Black men of all backgrounds (sexual, economic, and family), and (3) improve parent and adolescent relationships and communication.
  Arms: Waitlist Control

SUMMARY:
This study will develop and test the efficacy of an online, family-based intervention (MySTYLE) tailored to the relevant sexual health needs of non-heterosexual adolescent males and their parents/caregivers compared waitlist control group. Adolescent males and their parents will be recruited from community organizations, medical clinics and schools in Jackson, MS. Interviews with youth, parents, and relevant community leaders will inform the development of the interventions. Youth and their parents/caregivers in both intervention arms will complete three assessments in the four months after enrolling. This study will provide a wealth of information about the degree to which this intervention may be disseminated for this highly vulnerable population of young people.

DETAILED DESCRIPTION:
In recent years, the highest rates of HIV in the U.S. have been concentrated among young men who have sex with men (MSM), especially those of color. Unfortunately, evidenced-based intervention programs for non-heterosexual Black adolescent males (nHBAM) do not exist. Drs. Brown and Crosby have each designed, tested (in the context of NIH-funded RCTs) behavioral interventions targeting young people at-risk of HIV acquisition. Also, their previous work demonstrates that parental involvement prevents sexual risk behavior by adolescents. They will adapt key elements of STYLE, an efficacious HIV prevention program for adolescents and their parents/caregivers, to be relevant for nHBAM. A formative phase will use in-depth interviews to assess and identify the needs of nHBAM and their parents/caregivers. Work groups, composed of youth, parents/caregivers, stakeholders, and investigators, will tailor and refine the content in an iterative process with a sophisticated media company (MEE studios). MySTYLE is proposed to be a series of eight online novella episodes designed to increase relevant knowledge, attitudes, and sexual protective behaviors of nHBAM. The project will take place in Jackson MS, which has the highest prevalence of HIV among urban MSM in the U.S. and the third highest rate among Black MSM under the age of 25. Adolescents and parents will be recruited from community organizations, medical clinics and schools. The feasibility and effect sizes of MySTYLE, compared to a waitlist control group, will be tested with a cohort of 72 nHBAM and their parents. Interventions effect sizes will be determined for sexual behaviors, HIV testing, and psychosocial mediators (e.g., knowledge, attitudes, communication between adolescents and their parents/caregivers relative to sex, safer sex, and sexuality).

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for adolescents in all phases of the project will be: 1) at least 14 years of age but no more than 20; 2) stably-housed (have resided with the same adult caregiver for the past 6 months and no plans to leave the city or caregiver in the next 6 months). We understand that this will preclude homeless youth who may be at risk for HIV but MySTYLE will not be designed to address the numerous structural need of chronically homeless youth; 3) the ability to read and speak English; 4) identify as a biological male; 5) and identify racially as Black African American.

Eligibility criteria for Parents/caregivers for all phases of the project will be: 1) parent/caregiver or trusted adult of an adolescent who is potentially eligible for enrollment into the study; and 2) English speaking.

-

Exclusion Criteria: Exclusion criteria will be: a) not able to provide meaningful assent as determined by research staff, b) known HIV-infection (staff will facilitate entry into care if needed). Although we expect that most enrolled youth with be non-heterosexual Black adolescent males, heterosexual youth who enroll will be able to complete all intervention activities.

-

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescents must identify as biological male. Parent/caregiver may be male or female.
Enrollment: 72 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a dyad study. Adolescent participants were given the opportunity to invite a trusted adult to join them in the study; however, having a parent/guardian/trusted adult enroll was not mandatory. Only 7 trusted adults were enrolled. All enrollment values below indicate number of dyads, not individuals, unless otherwise stated.
Period: Overall Study
Arm/Group | MySTYLE | Waitlist Control
Started (Started: individuals - 46 MySTYLE, 33 Control) | 41 | 31
2 Month Follow-up (2 Month Follow-up: individuals- 27 MySTYLE, 28 Control) | 24 | 26
Completed (Completed: Individuals- 27 MySTYLE, 27 Control) | 23 | 25
Not Completed | 18 | 6
Not completed — Lost to Follow-up | 18 | 6

BASELINE CHARACTERISTICS:
Population: Notes: Baseline data is missing for one Waitlist Control Trusted Adult.
Groups:
- MySTYLE Adolescents; MySTYLE Trusted Adults: MySTYLE is online, brief and encourages parent-adolescent communication about sex and HIV prevention. Participants (non-heterosexual Black adolescent males and parents/caregivers) will receive two texts per week (for eight weeks) with links to intervention content that includes video, games and graphics to improve knowledge, motivation and skills for HIV prevention. Topics include assertive communication, sexual safety, goal setting, and resilience.
  MySTYLE: Youth and parents will receive two secure texts or emails to their cell phone or preferred device weekly (for eight weeks). Each text/email will contain a link to new media content designed to (1) improve sexual health knowledge surrounding HIV/AIDs and sexually transmitted infections, (2) increase acceptance of young Black men of all backgrounds (sexual, economic, and family), and (3) improve parent and adolescent relationships and communication.
- Waitlist Control Adolescents; Waitlist Control Trusted Adults: Participants randomized to the waitlist control will be eligible to receive the eight-week MySTYLE intervention after the completion of the 4-month follow-up assessment. During their first four months of participation, waitlist control participants will not receive any intervention materials.
  Waitlist Control: Youth and parents will not receive intervention materials for the first four months of participation. At the completion of the 4-month follow-up assessment, youth and parents will be eligible to receive two secure texts or emails to their cell phone or preferred device weekly (for eight weeks). Each text/email will contain a link to new media content designed to (1) improve sexual health knowledge surrounding HIV/AIDs and sexually transmitted infections, (2) increase acceptance of young Black men of all backgrounds (sexual, economic, and family), and (3) improve parent and adolescent relationships and communication.
- Total: Total of all reporting groups
Arm/Group | MySTYLE Adolescents | Waitlist Control Adolescents | MySTYLE Trusted Adults | Waitlist Control Trusted Adults | Total
Number analyzed (Participants) | 41 | 31 | 5 | 1 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (1.7) | 18.4 (1.5) | 38.0 (12.6) | 44.0 (NA) — only 1 participant | 18.2 (1.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/Gender Identity, customized
  Participants
    Male | 38 | 31 | 1 | 0 | 70
    Female | 1 | 0 | 4 | 0 | 5
    Trans male/trans man | 1 | 0 | 0 | 1 | 2
    Genderqueer/non-comforming | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at Birth Reported as female or male.
  Participants
    Female | 1 | 0 | 4 | 1 | 6
    Male | 40 | 31 | 1 | 0 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 41 | 30 | 5 | 1 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 39 | 28 | 4 | 1 | 72
  White | 0 | 0 | 1 | 0 | 1
  More than one race | 2 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Most Recent Grade Completed [Count of Participants; unit: Participants] — Population: Only adolescents, and not parents/caregivers, were asked this question. One waitlist control adolescent is missing data on this variable; therefore, only 30 were analyzed from this groups' 31 participants.
  Participants
    8th grade: number analyzed (Participants) | 41 | 30 | 0 | 0 | 71
    8th grade | 0 | 1 |  |  | 1
    9th grade: number analyzed (Participants) | 41 | 30 | 0 | 0 | 71
    9th grade | 1 | 1 |  |  | 2
    10th grade: number analyzed (Participants) | 41 | 30 | 0 | 0 | 71
    10th grade | 6 | 2 |  |  | 8
    11th grade: number analyzed (Participants) | 41 | 30 | 0 | 0 | 71
    11th grade | 3 | 1 |  |  | 4
    12th grade: number analyzed (Participants) | 41 | 30 | 0 | 0 | 71
    12th grade | 4 | 3 |  |  | 7
    Other: number analyzed (Participants) | 41 | 30 | 0 | 0 | 71
    Other | 27 | 22 |  |  | 49
Sexual Orientation [Count of Participants; unit: Participants] — Self-identified sexual orientation Population: Adults were not asked this question.
  Participants
    Exploring: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    Exploring | 3 | 2 |  |  | 5
    Undecided: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    Undecided | 1 | 1 |  |  | 2
    Questioning: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    Questioning | 2 | 0 |  |  | 2
    Other: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    Other | 1 | 0 |  |  | 1
    Gay: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    Gay | 16 | 16 |  |  | 32
    Bisexual: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    Bisexual | 6 | 4 |  |  | 10
    More than one endorsement: number analyzed (Participants) | 41 | 31 | 0 | 0 | 72
    More than one endorsement | 12 | 8 |  |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of an HIV Test at Study Completion
Description: Behavioral outcome: acceptance of a rapid, point of care HIV test at study completion. This will be assessed via electronic medical chart extraction.
Time Frame: 4 months post-baseline
Population: Missing data and those lost to follow-up account for the discrepancy in the analysis population. Only adolescent participants were offered an HIV test at study completion and analyzed on this outcome (no parent/caregivers).
Measure: Count of Participants; unit: Participants
Arm/Group | MySTYLE | Waitlist Control
Number analyzed (Participants) | 17 | 18
Participants
  No | 8 | 8
  Yes | 9 | 10

2. Primary Outcome: Change in Number of Condomless Anal Sex Acts at 4 Months
Description: Participants will be asked to report the number of condomless anal sex acts they have engaged in, in the past 90 days at baseline and at the 4 month follow-up. The change in number of condomless sex acts will be assessed.
Time Frame: 4-months post-baseline
Population: Only adolescents who completed the 4 month follow-up assessment were included.
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | MySTYLE Adolescents | Waitlist Control Adolescents | MySTYLE Trusted Adults | Waitlist Control Trusted Adults
Number analyzed (Participants) | 23 | 24 | 0 | 0
condomless anal sex acts | 0.7 (0.5) | 0.5 (0.8) |  |

3. Secondary Outcome: HIV Knowledge (Adolescent) at 4 Months
Description: The HIV Knowledge Scale assesses knowledge about issues such as risks for HIV, using 5 items with "true," "false," or "do not know" response options. Total scores range from 0 to 5. Higher scores indicate greater knowledge.
Time Frame: 4-months post-baseline
Population: Missing data and lost to follow-up account for the discrepancy in the analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MySTYLE | Waitlist Control
Number analyzed (Participants) | 23 | 24
score on a scale | 3.4 (0.8) | 3.5 (1.1)

4. Secondary Outcome: Parent Adolescent Sexual Communication Scale
Description: The Miller Sexual Communication Scale assesses the process and content of sexual communication between parents and adolescents. Only adolescent participants, not parent/caregivers, were asked to complete this scale. Evidence supports internal consistencies between .65 and .86. Each item is rated on a Likert scale 1 (not true) to 7 (very true) with scale scores ranging from 6-42. Higher scores indicate better communication about sexual behaviors.
Time Frame: Baseline, 2- and 4-months post-baseline
Population: Adolescents who completed 4 month follow-up assessment are analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MySTYLE Adolescents | Waitlist Control Adolescents | MySTYLE Trusted Adults | Waitlist Control Trusted Adults
Number analyzed (Participants) | 23 | 24 | 0 | 0
score on a scale | 20.1 (8.8) | 23.6 (9.5) |  |

ADVERSE EVENTS:
Time Frame: Data on adverse effects was collection from time of enrollment to end of follow-up, 4-months post-baseline.
Description: Adverse events as described in the study protocol were reported by study staff to the principle investigator.
Arm/Group | MySTYLE Adolescents | Waitlist Control Adolescents | MySTYLE Trusted Adults | Waitlist Control Trusted Adults
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/31 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/31 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/41 | 0/31 | 0/5 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03487796/Prot_SAP_000.pdf